CLINICAL TRIAL: NCT00588575
Title: In-Vivo Raman Spectroscopy of Barrett's Esophagus
Brief Title: Ramanspectroscopy in Barrett's Esophagus
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Louis-Michel Wong Kee Song, Principal Investigator, Mayo Clinic
Other Study IDs: 1999-04 00; DK67148; Raman
Record Dates: First submitted 2007-12-22; First posted 2008-01-08 (Estimated); Last update posted 2019-12-11 (Actual); Status verified 2009-09

CONDITIONS: Barrett's Esophagus
Keywords: Barrett's Esophagus
MeSH Terms: conditions — Barrett Esophagus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — esophageal biopsy
Oversight: Data Monitoring Committee: No

SUMMARY:
This study is being done to see if a new device, called near-infrared Raman spectroscopy, can provide similar information as that obtained from taking biopsies of the lining of your Barrett's esophagus

DETAILED DESCRIPTION:
In the search for means to enhance the surveillance of BE, optical spectroscopy is emerging as a candidate with high potential. Optical spectroscopic techniques measure specific light-tissue interactions, such as fluorescence, elastic scattering, and Raman (inelastic) scattering, which provide objective and quantitative diagnostic information about the molecular and/or structural status of tissue. Moreover, optical spectroscopy has the capacity to identify tissue pathology in situ in a rapid and non-destructive fashion. Among the optical spectroscopic techniques, near-infrared Raman spectroscopy (NIRS) is particularly promising because of the wealth of molecular-specific information contained in its spectra

ELIGIBILITY:
Inclusion Criteria:

* Closed to further enrollment

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Barrett's esophagus surveillance
Sampling Method: Non-Probability Sample
Enrollment: 119 (Actual)
Dates: Start 2004-10; Primary Completion 2007-05 (Actual); Study Completion 2007-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Louis M Wongkeesong, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States